CLINICAL TRIAL: NCT02510209
Title: Evaluation of the Teen Outreach Program in Hennepin County, Minnesota: Findings From the Replication of an Evidence-Based Teen Pregnancy Prevention Program
Brief Title: Evaluation of the Teen Outreach Program in Hennepin County, Minnesota
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abt Associates (Industry)
Collaborators: Hennepin County Human Services and Public Health Department (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TP1AH000078
Record Dates: First submitted 2015-07-27; First posted 2015-07-29 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Sexual Behavior; Pregnancy Early
Keywords: Teen pregnancy
MeSH Terms: conditions — Sexual Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Teen Outreach Program (Experimental)
  Interventions: Behavioral: Teen Outreach Program
- Control (No Intervention): Business as usual.

INTERVENTIONS:
Behavioral: Teen Outreach Program — TOP® is a youth development and service learning program for youth ages 12 to 17 designed to reduce teenage pregnancy and increase school success by helping youth develop a positive self-image, life management skills, and realistic goals. The TOP® program model consists of three components implemented in school, after school, or in community settings over nine consecutive months: (1) weekly curriculum sessions, (2) community service learning (CSL), and (3) positive adult guidance and support. The TOP® Changing Scenes® curriculum is separated into four age- and stage-appropriate levels, which range from Level 1, typically for youth ages 12 or 13, to Level 4, typically for youth age 17.
  Arms: Teen Outreach Program

SUMMARY:
This study tested the extent to which TOP®, when replicated with fidelity, produced impacts on sexual risk-taking behaviors in the short term and the longer term.

DETAILED DESCRIPTION:
This is a cluster randomized controlled trial. Teachers were randomized within schools to the treatment and control conditions. To assess the impact of offering TOP®, students were surveyed three times: at baseline, before the intervention began for the treatment group; 12 months after baseline (short-term impacts); and 24 months after baseline (long-term impacts). Baseline data and subsequent follow-up data were collected using a Web-based survey. Paper surveys were used as back-up for baseline data collection. The pooled survey data from two school-year cohorts (school years 2011-2012 and 2012-2013) were used to estimate program impacts using an intent-to-treat (ITT) analysis. Program fidelity and interview data were used to describe program implementation.TOP® was delivered in middle schools, high schools, alternative schools, and public charter schools in Hennepin County. It was implemented during school hours in classes that spanned an entire school year with the same cohort of students. The subject of the class in which TOP® was placed differed across schools (for example, social studies, study hall, health).

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in a study teacher's class at the time of the baseline survey
* Active parental consent and youth assent

Exclusion Criteria:

* Inability to complete survey in the languages provided
* Prior participation in TOP

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1644 (Actual)
Dates: Start 2011-07; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Sex in the last 90 days | 12 months after baseline
  Single dichotomous item on self-report questionnaire

SECONDARY OUTCOMES:
Sex without contraception in the last 90 days | 12 months after baseline
  Single dichotomous item on self-report questionnaire
Sex in the last 90 days | 24 months after baseline
  Single dichotomous item on self-report questionnaire
Sex without contraception in the last 90 days | 24 months after baseline
  Single dichotomous item on self-report questionnaire
Ever had sex | 12 months after baseline
  This outcome was measured among the subgroup of participants who had never had sex at baseline. Single dichotomous item on self-report questionnaire.
Ever had sex | 24 months after baseline
  This outcome was measured among the subgroup of participants who had never had sex at baseline. Single dichotomous item on self-report questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Francis, PhD, Study Director — Abt Associates Inc.
Locations (1):
- Hennepin County Human Services and Public Health Department, Minneapolis, Minnesota, United States

REFERENCES:
- [Result] Francis, K., Woodford, M., and Kelsey, M. (2015). "Evaluation of the Teen Outreach Program in Hennepin County, MN: Findings from the Replication of an Evidence-Based Teen Pregnancy Prevention Program." Cambridge, MA: Abt Associates Inc.